CLINICAL TRIAL: NCT00258765
Title: A Phase IIb Randomised Clinical Trial of the Tolerability, Safety and Efficacy of Adjuvant Docetaxel-Zoledronic Acid After Prostatectomy for High-risk Early Prostate Cancer (AD-ZAP).
Brief Title: Adjuvant Docetaxel-Zoledronic Acid in High-risk Early Prostate Cancer Following Prostatectomy.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment & not feasible to continue
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CZOL446GAU15
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Prostate Cancer
Keywords: zoledronic acid; prostate cancer; high risk; PSA; docetaxel
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoledronic Acid (Experimental)
  Interventions: Drug: Zoledronic Acid
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Zoledronic Acid
  Arms: Zoledronic Acid
Drug: Docetaxel
  Arms: Docetaxel

SUMMARY:
Radical prostatectomy is used to treat early prostate cancer in otherwise well men, but is followed by later cancer relapse in 1 in 4 cases. This study aims to see if post-operative adjuvant therapy with a combination of zoledronic acid and docetaxel might help reduce relapse in such cases. Patients will be randomized to receive the adjuvant combination therapy or no therapy. All patients will be monitored closely for signs of relapse and treated appropriately with conventional salvage therapy.

ELIGIBILITY:
Inclusion Criteria:

* Radical prostatectomy for prostate cancer within last 2 months.
* Post-operative Kattan nomogram predicts >25% risk of PSA relapse by 5 years.
* 6-week post-operative serum PSA<0.2ng/mL.
* Low levels of circulating prostate cancer cells in the blood, detected by PCR amplification of PSA mRNA 6 weeks post-prostatectomy.

Exclusion Criteria:

* Pre-operative serum PSA level >20ng/ml.
* Clinical evidence of metastases by 6-week post-operative visit.
* Prior treatment with either ADT or bisphosphonate therapy.
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g.extraction, implants)

Other protocol defined inclusion / exclusion criteria may apply.

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-05; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
safety and tolerabilty of adjuvant chemotherapy with docetaxel and Zometa | 6 months after study entry

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Sydney, Australia

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=717